CLINICAL TRIAL: NCT06240481
Title: Study to Assess the Efficacy of Two Brushing Regimens in the Reduction of Dental Plaque and Aid of Gum Problems
Brief Title: Clinical Research Study to Assess the Efficacy of Two Brushing Regimens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2024-02-PG-MRG-SP-BGS
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-01

CONDITIONS: Dental Plaque; Gingivitis
Keywords: plaque; gingivitis; Loe and Silness Gingival Index; Quigley and Hein Plaque Index
MeSH Terms: conditions — Dental Plaque; Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Meridol regimen comprises an amine base compound, zinc lactate and NaF (AZF) toothpaste and mouthwash, brush 2x day/2min and swish 15ml/30 secs after brushing
  Interventions: Drug: Test Regimen; Drug: Control Regimen
- Group II (Placebo Comparator): Regular fluoride toothpaste, Brush 2 x day 2 mins
  Interventions: Drug: Test Regimen; Drug: Control Regimen

INTERVENTIONS:
Drug: Test Regimen — toothpaste & mouthwash
Drug: Control Regimen — toothpaste

SUMMARY:
The objective of this twelve-week clinical research study is to assess the efficacy of two brushing regimens: 1) toothpaste with mouthwash containing sodium fluoride/zinc and manual toothbrush as compared to 2) regular fluoride toothpaste and manual toothbrush in the reduction of dental plaque and aid of gum problems.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects aged 18-70 years, inclusive.
* Availability for the twelve-week duration of the clinical research study.
* Good general health based on the opinion of the study investigator
* Minimum of 20 permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification)

Exclusion Criteria:

* Presence of orthodontic appliances.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Moderate and/or advanced periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study.
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study. -Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients. -On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating and/or drinking for periods up to 4 hours.
* History of alcohol and/or drug abuse.
* Self-reported pregnancy and/or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Quigley and Hein Plaque Index | Baseline, 3 weeks, 6 week & 12 weeks
  reductions in dental plaque
Loe and Silness Gingival Index | Baseline, 3 weeks, 6 week & 12 weeks
  assessment of gum problems (gingival scores)

CONTACTS AND LOCATIONS:
Overall Officials: Augusto R Elias-Boneta, DMD, MSD, Principal Investigator — Clinica Dental Dr. Sitges Carretera de Cardona
Locations (1):
- Clinica Dental Dr. Sitges, Manresa, Spain

IPD SHARING:
Plan to Share IPD: No